CLINICAL TRIAL: NCT06427213
Title: A Study of the Zanubrutinib-containing Regimens in Patients With Newly Diagnosed Mantle Cell Lymphoma
Brief Title: This is a Phase II, Open-label, Multicentre Study of Zanubrutinib-containing Regimens in Patients With Newly Diagnosed Mantle Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-TN MCL
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-01

CONDITIONS: Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin
Keywords: Zanubrutinib
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — zanubrutinib; obinutuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elder Patients（≥65） (Experimental): Induction: Zanubrutinib and Obinutuzumab 1year
  Maintenance: Zanubrutinib continued until progression
  Interventions: Drug: Zanubrutinib,Obinutuzumab
- Young Patients with High risk （≥18，<65） (Experimental): Induction: Zanubrutinib and R-BAC 6 cycles
  Consolidation: ASCT（If eligible for transplantation），Otherwise, the patient was directly entered into maintenance treatment
  Maintenance: Zanubrutinib continued until progression
  Interventions: Drug: Zanubrutinib and R-BAC

INTERVENTIONS:
Drug: Zanubrutinib,Obinutuzumab — Zanubrutinib, 160mg PO BID. C1D17 continuously for 1 year or until progressive disease； Obinutuzumab ：Obinutuzumab will be administered 1,000 mg intravenously on days 1, 8, and 15 of cycle 1, then 1,000 mg on day 1 of cycles 2 to 6, then 1,000 mg every 8 weeks，up to 20 doses. 1 cycle = 28 days.
  Maintenance: Zanubrutinib, 160mg PO BID
  Arms: Elder Patients（≥65）
Drug: Zanubrutinib and R-BAC — Induction: Zanubrutinib and R-BAC 6 cycles
  Consolidation: ASCT（If eligible for transplantation），Otherwise, the patient was directly entered into maintenance treatment
  Maintenance: Zanubrutinib continued until progression
  Arms: Young Patients with High risk （≥18，<65）

SUMMARY:
This is a phase II, open-label, multicentre study of Zanubrutinib-containing regimens in patients with newly diagnosed mantle cell lymphoma.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, investigator-initiated clinical trial to evaluate the efficacy and safety of zanubrutinib-containing regimens in the treatment of newly diagnosed elderly or young patients with high risk MCL, aiming to find a more optimal treatment regimen for elderly or young patients with high risk MCL to improve the efficacy, survival time and quality of life of patients.

In elderly patients arm：patients start with the induction therapy of zanubrutinib combined with obinutuzumab for 1 year and then entered the maintenance therapy of zanubrutinib orally until intolerable toxicity or disease progression

In young patients with high risk arm：patiens <65 years，and meet one or more of the following risk factors: TP53 mutation, blastoid/pleomorphic type, high sMIPI score. patients start with 6 cycles of induction therapy with zanubrutinib combined with R-BAC regimen, and the patients who achieve CR/PR and meet the transplantation criteria will receive ASCT consolidationand, then received maintenance therapy with zanubrutinib. otherwise, Patients who is ineligible for transplantation，will take zanubrutinib orally until intolerable toxicity or disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in clinical study; Fully understand and understand the study and sign the informed consent form (ICF);Willingness to follow and ability to complete all study steps
2. Histopathologically confirmed mantle cell lymphoma according to the 5th edition of the World Health Organization (WHO)，previous untreatment for mantle-cell lymphoma (MCL)
3. The elderly group ≥65 years old;The young group was ≥18 years old and < 65 years old.
4. ECOG Performance Status 0-3
5. Life expectancy of at least 3 months
6. At least one evaluable lesion according to 2014 Lugano criteria;
7. Proper functioning of the major organs, no major heart, lung, liver, kidney, or immunodeficiency (no blood transfusion, granulocyte colony-stimulating factor, or other medical support within 7 days before starting the study) :Hemoglobin (HB)≥60 g/L;Absolute neutrophil count(ANC)≥0.5×10^9/L;Platelet count（PLT）≥50×10^9/L;AST and ALT ≤ 2.5 x ULN；Total bilirubin ≤ 1.5 times the ULN;Ccr≥40ml/min（Cockcroft-Gault ）；Left Ventricular Ejection Fraction (LVEF) ≥ 50%

Exclusion Criteria:

1. The presence of other tumors could affect the study medication or interfere with the results;
2. Patients require treatment with strong or moderate CYP3A inhibitors;
3. Pregnant or lactating women;
4. Known to be allergic to the test drug ingredients;
5. Subjects of childbearing potential who are unwilling to use highly effective contraceptive methods;
6. Live vaccination was administered within 28 days prior to treatment
7. Known human immunodeficiency virus (HIV) infection or suggested active B or C infection The following serologic status of hepatitis C virus infection: 1) Hepatitis B virus (HBV) DNA positive. Positive hepatitis B surface antigen (HBsAg) or anti-hepatitis B core antibody (HBcAb) seropositive if HBV DNA is undetectable and willing to accept Monthly surveillance for HBV reactivation was eligible. 2) Hepatitis C virus (HCV) antibody positive. For patients with HCV antibodies present, if undetectable HCV RNA, can be included;
8. Severe coagulopathy and serious impairment of heart, brain, lung, liver, kidney and other organs
9. History of deep vein thrombosis (DVT) or pulmonary embolism (PE) within the past 12 months;
10. Any risk that is considered by the investigator to be likely to affect the safety of the subjects or to pose a risk to the study And vital diseases, medical conditions, or organ system insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response rate after induction | 3 yeas
  Objective Response rate will be determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Complete remission rate after Interim treatment | 3 years
  Complete remission rate will be determined on the basis of investigator assessments according to 2014 Lugano criteria.
MRD negativity rate after induction | 3 years
  MRD negativity rate after induction treatment
Progression free survival (PFS) | 5 years
  The time from start of treatment to progression or death from any cause
Overall survival (OS) | 5 years
  The time from start of treatment to death from any cause
Percentage of Participants With Adverse Events | 5 years
  Adverse Events will be determined and graded on the basis of investigator assessments according to NCI CTC AE 5.0